CLINICAL TRIAL: NCT05046028
Title: Individual Nutritional Support With High Protein Formula With Modified Sensory Component for H&N Cancer Patients on Chemo and Radiotherapy
Brief Title: Individualization of Nutritive Sensory Support Of Radiation Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Gevorkov Artem R, senior researcher, radiotherapist, National Medical Research Radiological Centre of the Ministry of Health of Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INSSORT
Record Dates: First submitted 2021-06-02; First posted 2021-09-16 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Radiotherapy; Complications; Head and Neck Cancer
Keywords: Nutritional support; Radiotherapy; Head and Neck Cancer; Complications
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Dietary Supplements; Taste

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): 50 patients with squamous cell head cancer over 18 years of age, receiving chemoradiation therapy, receiving 3 bottles (х 200 ml) of ONS with Protein Oncosensation with a neutral taste throughout the course of treatment.
  Interventions: Dietary Supplement: Oral nutritional supplements (ONS) with a cooling effect + ONS without a sensor component and taste + standard diet
- Prospective Control group (Active Comparator): 50 patients over 18 years of age with squamous cell carcinoma of the head and neck, receiving chemoradiation therapy, receiving standard nutritional therapy with a neutral taste throughout the course of treatment.
  Interventions: Dietary Supplement: ONS without a sensor component and taste + standard diet
- Retrospective Control group (Sham Comparator): 60 patients who received chemoradiotherapy earlier with standard nutritional support.
  Interventions: Dietary Supplement: Standard diet

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplements (ONS) with a cooling effect + ONS without a sensor component and taste + standard diet — ONS with a cooling effect and Red Fruits taste. 3 bottles (х 200 ml) per day X 14 days (at severe mucositis period) in addition to a standard diet and other ONS without a sensor component and taste according to protein and energy requirements based on ESPEN guidelines (protein 1.5 g/kg/day and Energy -25 and 30 kcal/kg/day)
  Arms: Test
Dietary Supplement: ONS without a sensor component and taste + standard diet — Nutritional support + ONS without a sensor component and taste (cooling effect) in addition to a standard diet according to protein and energy requirements based on ESPEN guidelines (protein 1.5 g/kg/day and Energy -25 and 30 kcal/kg/day)
  Arms: Prospective Control group
Dietary Supplement: Standard diet — Without appropriate nutritional support - not in accordance with current ESPEN guidelines (protein and Energy intake less than 1.5 g/kg/day and 25 and 30 kcal/kg/day). (Historical retrospective control).
  Arms: Retrospective Control group

SUMMARY:
Nutritional deficiency and subsequent weight loss in patients with head and neck cancer is a common problem and a negative predictor of treatment outcomes and mortality, as well as quality of life. Nutritional support for patients is a prerequisite for the successful management of cancer patients. Sensory changes can be side effects of chemotherapy or ionizing radiation, which damages sensory receptors in the area of radiation, disrupts the function of the salivary glands, leading to hyposalivation and a decrease in taste. Individual choice of nutrition based on sensory sensations can significantly improve the quality of life of patients and ensure timely correction of their eating behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* The presence of morphological verification of squamous cell carcinoma of the head and neck
* No history of anticancer treatment
* ECOG score 0 - 2
* Life expectancy is more than 3 months
* Normal liver, kidney and bone marrow function
* Absence of severe uncontrolled concomitant chronic diseases and acute diseases (including infectious diseases)
* Absence of pregnancy, lactation
* Initial compliance of patients (according to the consultation of a psychologist and questionnaires) with a signed informed consent

Exclusion Criteria:

* Simultaneous participation in another clinical trial
* Failure to meet inclusion criteria
* The patient's condition is ECOG ≥3, Karnovsky ≤40%.
* Bleeding
* Decay / Abscess in the area of tumor lesion
* Pregnancy or breastfeeding
* Refractory cachexia
* Allergy or intolerance to any of the components of ONS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | 1 year
  QoL is evaluated and recorded according to questionnaire The Functional Assessment of Cancer Therapy - Fatigue (FACT-F)
Nutritional status | 1 year
  Nutritional status is evaluated and recorded according to Nutritional Risk Screening (NRS) 2002
Patient compliance | 1 year
  The level of patient compliance is evaluated and recorded according to Morisky 8-Item Medication Adherence Questionnaire.

SECONDARY OUTCOMES:
Tolerance to chemoradiation therapy - mucositis | 4 months
  Mucositis as adverse event of chemoradiation therapy is evaluated and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Tolerance to chemoradiation therapy - dermatitis | 4 months
  Dermatitis as adverse event of chemoradiation therapy is evaluated and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Terms of treatment | during radiation treatment
  Terms of treatment is recorded in total number of days from the first day of radiation treatment to the last one.
Unplanned breaks | during radiation treatment
  Days of delayed treatment
Efficiency of chemoradiation therapy | 1 year
  Degree of tumor resorption by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
1-year locoregional control | 1 year
  1-year locoregional control after chemoradiation therapy
1-year overall survival | 1 year
  1-year overall survival is the percentage of people who are alive one year after they started chemoradiation therapy
1-year relapse-free survival | 1 year
  1-year relapse-free survival is the percentage of people who have not had relaps one year after they started chemoradiation therapy
Dynamics of sensory changes | 1 year
  Dynamics of sensory changes based on the adapted total soluble solids scale (TSS scale)
Dynamics of pain syndrome | 1 year
  Dynamics of pain syndrome based on numerical rating scale (NRS scale)

CONTACTS AND LOCATIONS:
Locations (1):
- P. Hertsen Moscow Oncology Research Institute, Moscow, Russia